CLINICAL TRIAL: NCT05675189
Title: An In Depth Study Examining Patterns in the Clinical Trial Experiences of Migraine Patients
Brief Title: Exploring Clinical Trial Experiences of Patients With Migraine
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 81287400
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Migraine; Migraine Disorders
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation has historically been heavily biased toward specific demographics.

This study will invite several participants to gather a wide range of information on clinical trial experiences for migraine patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of migraine.

People with migraine who are invited to take part in medical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a minimum of 18 years of age
* Patient has been diagnosed with a type of migraine
* Patient plans to participate in an interventional clinical trial for the condition of migraine
* Patient has access to a home internet connection in order to provide regular updates through the course of the study

Exclusion Criteria:

* Patient has an ECOG score of 4 or higher
* Patient is not able to provide consistent digital updates as per study requirements
* Patient does not complete or agree to terms outlined in the Informed Consent Form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with migraine who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a migraine clinical trial | 3 months
Rate of patients who remain in migraine clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peters GL. Migraine overview and summary of current and emerging treatment options. Am J Manag Care. 2019 Jan;25(2 Suppl):S23-S34. PMID 30681821
- [Background] Tfelt-Hansen P. Understanding clinical trials in migraine. J Headache Pain. 2006 Apr;7(2):101-8. doi: 10.1007/s10194-006-0278-2. Epub 2006 Mar 31. PMID 16575501
- [Background] Solomon S. Selection of patients for clinical drug trials in migraine. Neuroepidemiology. 1987;6(4):164-71. doi: 10.1159/000110115. PMID 3317096

DOCUMENTS (1):
  • Informed Consent Form (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT05675189/ICF_000.pdf